CLINICAL TRIAL: NCT00086164
Title: A Phase 1/2, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Pilot Trial to Assess the Effect of Treatment of the Recipient Vein of a Polytetrafluoroethylene (PTFE) Vascular Access Graft With Two Concentrations of E2F Decoy as Compared to Placebo on Neointimal Hyperplasia and the Preservation of Graft Function in Patients With Chronic Renal Failure Requiring Hemodialysis
Brief Title: Prevention of Vascular Access Graft Failure in Patients With Chronic Renal Failure Requiring Hemodialysis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Anesiva, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: CGT003-05
Record Dates: First submitted 2004-06-25; First posted 2004-06-29 (Estimated); Last update posted 2005-07-19 (Estimated); Status verified 2005-07

CONDITIONS: Hyperplasia; Chronic Renal Failure
Keywords: edifoligide; E2F Decoy; Chronic Renal failure; hemodialysis; AV Graft; neointimal hyperplasia
MeSH Terms: conditions — Hyperplasia; Kidney Failure, Chronic | interventions — edifoligide

INTERVENTIONS:
Drug: edifoligide (E2F Decoy)

SUMMARY:
The purpose of this study is to determine the effect of recipient vein pretreatment of edifoligide (E2F Decoy), compared to placebo, on graft/recipient vein stenosis in polytetrafluoroethylene (PTFE) vascular access grafts placed for hemodialysis at 6 months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Be scheduled to undergo placement of a new straight or loop arm PTFE arteriovenous hemodialysis access graft or a Vectragraft® (Thoratec, Inc.)
* Be currently receiving chronic dialysis or be expected to begin hemodialysis within 4 weeks of placement of the index PTFE graft
* Have undergone an assessment of patency (such as venography) of central veins if any of the following conditions have occurred on the ipsilateral arm intended for graft placement: presence of collateral veins, upper extremity edema or increased size (relative to the contralateral arm), history of subclavian catheter, transvenous pacemaker, or history of trauma or surgery that may have involved the neck or chest veins
* Be > 18 and <80 years old
* Have a documented negative serum pregnancy test (for all women of childbearing potential)
* Be using an acceptable method of birth control if of reproductive potential and agree to continue using the birth control for at least 3 months following the graft procedure
* Have agreed to participate voluntarily and have signed and dated an IRB/EC approved, Patient Informed Consent form

Exclusion Criteria:

* Have an intended recipient vein >6 mm or <3 mm in diameter
* Have a history of three or more previous PTFE grafts
* Have uncorrected central vein (including the subclavian vein) stenosis
* Have markedly diminished arterial pulses in the access location (unless adequate flow has been documented by arteriography or Doppler ultrasound)
* Anticipate receipt of a renal transplant within 6 months of enrollment into this study
* Have anticipated use of the index PTFE graft <14 days after enrollment (this does not apply to Vectragraft®)
* Have a known allergy to iodinated contrast
* Have a known hypercoagulable state (e.g., antithrombin III deficiency; antiphospholipid or anticardiolipin antibodies; Factor V Leiden; circulating lupus anticoagulant; current, active, heparin-induced thrombocytopenia; Protein C or S deficiency; or a history of recurrent deep venous thrombosis not related to AV access)
* Have been in another investigational (i.e., nonapproved) drug or device study within the previous 30 days or prior participation in another clinical study with E2F Decoy
* Have been previously enrolled in this study for an earlier access graft
* Have any comorbid, nonrenal condition that makes 6-month survival questionable (e.g., end-stage cancer, advanced heart failure)
* Have a known or suspected history of drug or alcohol abuse within the previous 6 months
* Have a known allergy to any component of the investigational product (drug or device), including latex

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-05

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - National Institute of Clinical Research, American Medical Tower, Los Angeles, California
  - Outcomes Research International, Inc., Hudson, Florida
  - University of Miami, School of Medicine, Miami, Florida
  - Tampa General Hospital, Tampa, Florida
  - LifeLink Transplant Institute, Tampa, Florida
  - Emory University, Renal Division, Atlanta, Georgia
  - University Transplant, Chicago, Illinois
  - Stoney Island Dialysis, Chicago, Illinois
  - Methodist Hospital, Tower Surgical, Indianapolis, Indiana
  - Vascular Surgery Associates, Baton Rouge, Louisiana
  - Tulane Center for Abdominal Transplant, New Orleans, Louisiana
  - Henry Ford Hospital, Detroit, Michigan
  - Thoracic & Cardiovascular Healthcare Foundation, Lansing, Michigan
  - St. Louis University, Division of Nephrology, St Louis, Missouri
  - NYU Medical Center, New York, New York
  - St. Luke's Hospital, Department of Surgery, New York, New York
  - University of Rochester, The Center for Vascular Disease, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Surgical Education, Greenville, South Carolina
  - University of Utah School of Medicine, Dept of Surgery, Salt Lake City, Utah
  - Nephrology Clinical Research Center, Charlottesville, Virginia